CLINICAL TRIAL: NCT02286193
Title: Creating a Clinic-Community Liaison Role in Primary Care: Engaging Patients and Community in Health Care Innovation
Acronym: LINCC
Status: Completed | Type: Observational
Sponsor: Kaiser Permanente (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 1011 Hsu PCORI Cycle 1
Record Dates: First submitted 2014-11-05; First posted 2014-11-07 (Estimated); Results first posted 2016-09-07 (Estimated); Last update posted 2017-11-13 (Actual); Status verified 2017-10

CONDITIONS: Patient Engagement; Community Integration
MeSH Terms: conditions — Patient Participation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients presenting to Community Resource Specialist (CRS): Primary care patients who are referred or self-refer to the CRS for education and linkage to community resources that can help support health goals
  Interventions: Behavioral: Patient clinical encounters with Community Resource Specialist (CRS)

INTERVENTIONS:
Behavioral: Patient clinical encounters with Community Resource Specialist (CRS) — CRS will work with patients to create goals, develop action plans and link to community resources to support goals

SUMMARY:
This project will engage patients and health care teams to develop, implement, and rigorously evaluate a new lay health worker role (Community Resource Specialist, CRS) for primary care teams. The CRS will link patients and healthcare clinics with community resources.

DETAILED DESCRIPTION:
Patients are served best when multiple organizations work together to meet healthcare needs. In the Chronic Care Model, community resources supplement productive interactions between patients and care teams. However, healthcare delivery systems and health research have given relatively little attention to the model's community features. This project engages patients in designing a primary care community liaison role (Community Resource Specialist, CRS) connecting patients to clinic and community resources that support chronic disease prevention and management. The CRS role will enhance primary care by better integrating community resources into patient care.

The proposed design effort will:

* develop tools and work processes that promote meaningful patient engagement in creating a CRS concept and role
* integrate the CRS role into primary care teams
* assess effects of this role on patient-centered outcomes.

The patient engagement process will use principles from Lean, a quality improvement method, to engage all primary care stakeholders, particularly patients and clinical staff. The project will integrate community resources into the patient-centered medical home model of Group Health, a nonprofit healthcare system that provides coverage and care.

The project will enhance patient resources and options for managing and preventing chronic illness and improve patient-centered outcomes.

The project's specific aims are:

* Aim 1: Develop, implement, and evaluate new methods to involve patients intensively in care design. The investigators will create processes and tools to select and train participants and facilitate their productive contributions to care design. The investigators will document the approach's benefits and challenges using qualitative and quantitative data.
* Aim 2: Design and pilot a new CRS role for primary care teams. Robust engagement of patients in designing this new primary care team role will result in innovative, patient-centered solutions. The investigators will pilot this service at three clinics. The aim of the new service is to help patients more readily access the healthcare and community resources they need for preventing and treating chronic disease. The CRS also may help educate clinic staff about available community resources and increase the primary care team's use of holistic approaches to health.
* Aim 3: Evaluate the design and efficacy of the CRS. The investigators will conduct both formative and outcome evaluations of the CRS role.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled at Group Health Cooperative, Seattle, Washington, in one of three pilot primary care clinics
* Referred or self-referred to the CRS for connection to community resources to support health goals

Exclusion Criteria:

* Not enrolled at Group Health
* Not enrolled in one of the pilot clinics

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Group Health primary care patients at one of three pilot clinics who are referred or self-refer to work with a Community Resource Specialist (CRS)
Sampling Method: Non-Probability Sample
Enrollment: 418 (Actual)
Dates: Start 2013-03; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clarissa Hsu, PhD, Principal Investigator — Group Health Research Institute

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment period was 15 months, from July 2014 - December 2015.
Pre-assignment Details: This was a single group observational study. All patients were considered enrolled who received care at one of 3 pilot clinics and were referred or self-referred to receive services from the Community Resource Specialist (CRS). They were considered "complete" if after referral they completed at least 1 phone or in-person CRS visit.
Period: Overall Study
Arm/Group | Patients Presenting to Community Resource Specialist (CRS)
Started | 622
Completed | 418
Not Completed | 204
Not completed — Referred: CRS unable to make contact | 62
Not completed — Referred: unable to reach/resource sent | 104
Not completed — Referred: Declined service | 38

BASELINE CHARACTERISTICS:
Arm/Group | Patients Presenting to Community Resource Specialist (CRS)
Number analyzed (Participants) | 418
Age, Customized [Number; unit: participants]
  Less than or equal to 18 | 70
  19 - 34 | 38
  35 - 64 | 165
  65 or older | 145
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 305
  Male | 113
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 12
  Asian | 49
  Black or African American | 83
  Native Hawaiian or Other Pacific Islander | 11
  White | 228
  Other | 20
  Unknown | 15

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Receiving a Resource for Community Services
Description: Number of patients who completed at least one visit with the CRS and were given a referral for at least one resource, service, or organization. This was assessed by abstraction and coding of CRS documentation in the medical record.
Time Frame: 3 months
Measure: Number; unit: participants
Groups:
- Patients Presenting to Community Liaison: Primary care patients who are referred or self-refer to the CRS for education and linkage to community resources that can help support health goals
Arm/Group | Patients Presenting to Community Liaison
Number analyzed (Participants) | 418
participants | 356

2. Secondary Outcome: Number of Participants Setting a Goal With Their CRS
Description: Number of patients who completed at least one visit with the CRS and set a specific action-based goal with their CRS. Patients could meet with the CRS and receive referrals to resources without setting specific action-based goals. This was assessed by abstraction and coding of CRS documentation in the medical record.
Time Frame: 3 months
Measure: Number; unit: participants
Arm/Group | Patients Presenting to Community Resource Specialist (CRS)
Number analyzed (Participants) | 418
participants | 162

ADVERSE EVENTS:
Description: No adverse events were reported to us. However this was not a clinical trial. It was an evaluation of a delivery system innovation.
Arm/Group | Patients Presenting to Community Resource Specialist (CRS)
Serious Adverse Events (participants affected / at risk) | 0/418
Other Adverse Events (participants affected / at risk) | 0/418

LIMITATIONS AND CAVEATS:
This was not a clinical trial. It is was a single-group observational evaluation of a delivery system innovation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No